CLINICAL TRIAL: NCT06954259
Title: Prognostic Correlation Between the Ratio of the Neutrophil Ratio to the Ratio of CD4+/CD8+ T Cells in Patients With Advanced Non-small Cell Lung Cancer NSCLC) Undergoing Immunotherapy Combined With Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Qiang Xu (Other)
Responsible Party: Sponsor-Investigator, Qiang Xu, Jiangxi Provincial Cancer Hospital, Jiangxi Provincial Cancer Hospital
Organization: Jiangxi Provincial Cancer Hospital (Other)
Other Study IDs: 2025ky010
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: NSCLC; lung cancer; pulmonary carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the prognostic correlation between the neutrophil ratio and the ratio of CD4+/CD8+ T cells in patients with advanced non-small cell lung cancer (NSCLC) who receive immunotherapy combined with chemotherapy, with the aim of providing references for clinical treatment.

DETAILED DESCRIPTION:
According to the content released in the Global Cancer Statistics Report 2022 (Global Cancer), lung cancer is the leading cause of cancer-related deaths worldwide. Traditional treatment methods such as surgery, radiotherapy, and chemotherapy have limitations in their curative effects. Immune checkpoint inhibitors (ICIs) have greatly changed the treatment landscape of non-small cell lung cancer (NSCLC). Although progress has been made in immunotherapy, the prediction of its efficacy relies on methods such as Tumor Mutational Burden (TMB) and the expression of PD-L1. Therefore, finding more effective treatment strategies and prognostic evaluation indicators has become a key task in lung cancer research. Relevant studies have delved into the prognostic and predictive values of inflammation-related peripheral blood biomarkers in NSCLC patients receiving immunotherapy. The Neutrophil-to-lymphocyte ratio (NLR) has emerged as a potential biomarker for cancer prognosis. However, lymphocyte subsets can be influenced by factors such as race, age, medications, gender, stress, physical activity, and lifestyle. In this study, CD4+/CD8+ T cells were selected to eliminate the influence of individual differences, and it is intended to investigate whether there is a prognostic correlation of CD4+/CD8+ T cells in the immunotherapy combined with chemotherapy for patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* (1)Inoperable stage III or IV NSCLC (AJCC 8th edition TNM staging) confirmed by pathological histology or cytology.(2)Received first - line immunotherapy (PD - 1/PD - L1 inhibitors) combined with chemotherapy, and driver genes are negative.(3)There is at least one measurable lesion in the lungs on CT imaging (RECIST 1.1).(4)Have complete clinical data.(5)The patient or the authorized family member gives informed consent.

Exclusion Criteria:

* (1)Have gene mutations such as EGFR/ALK/ROS1 and have not received standardized targeted therapy.(2)Have a second primary malignant tumor concurrently.(3)Have been infected or used antibiotics within 7 days before blood sampling.(4)Have severe abnormalities in the functions of organs such as the heart, liver, lungs, kidneys, and bone marrow.(5)Have other autoimmune diseases and endocrine and metabolic diseases concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC who received immunotherapy combined with chemotherapy at Jiangxi Provincial Cancer Hospital
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Remission Rate | Recruit patients with non-small cell lung cancer who received immunotherapy combined with chemotherapy from July 2022 to June 2024. Count the percentage of patients who achieved complete response or partial response, and the calculation deadline is April
  The objective response rate (ORR) is defined as the percentage of patients who achieve a complete response (CR) or a partial response (PR) among all the patients who have received the treatment.
Progression - Free Survival | Recruit patients with non-small cell lung cancer who received immunotherapy combined with chemotherapy from July 2022 to June 2024. Count the duration from the initiation of immunotherapy combined with chemotherapy to the date of the first documented dis
  The Progression-Free Survival (PFS) is defined as the duration from the initiation of immunotherapy combined with chemotherapy to the date of the first documented disease progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China